CLINICAL TRIAL: NCT02790957
Title: Effect of a Single Plerixafor Injection on Diabetic Wound Healing. A Pilot, Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Plerixafor in Diabetic Wound Healing
Acronym: MOZOBL07740
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety reasons
Sponsor: Gian Paolo Fadini (Other)
Collaborators: University Hospital Padova (Other)
Responsible Party: Sponsor-Investigator, Gian Paolo Fadini, Associate Professor, University of Padova
Organization: University of Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3694/Ao/15
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Diabetes; Wounds; Critical Limb Ischemia
MeSH Terms: conditions — Diabetes Mellitus; Wounds and Injuries; Chronic Limb-Threatening Ischemia | interventions — plerixafor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plerixafor (Experimental): Single subcutaneous injection of Plerixafor (0.24 mg/kg)
  Interventions: Drug: Plerixafor
- Placebo (Placebo Comparator): Single injection of an equal volume of NaCl solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Plerixafor — Single injection of 0.24 mg/kg Plerixafor
  Other Names: Mozobil
  Arms: Plerixafor
Drug: Placebo — Single injection of an equal volume of NaCl solution
  Arms: Placebo

SUMMARY:
Chronic non-healing wounds represent a major source of morbidity, disability, and mortality in diabetic patients. Diabetes is the leading cause of non-traumatic limb amputations worldwide. Many patients with ischemic or neuroischemic wounds are not candidate to surgical/endovascular revascularization, owing to anatomical vascular reasons or for the underlying conditions and co-morbidities. Therefore, identification of novel medical treatment strategies to improve wound healing in diabetic patients is a major challenge for clinicians, researchers, and health care systems.

Defects in bone marrow (BM)-derive stem and progenitor cells, including EPCs (endothelial progenitor cells), contribute to diabetic complications. Stem cell mobilizing agents have been previously studied as an adjunctive therapy for critical limb ischemia and chronic non-healing wounds in diabetic and non-diabetic patients, as well as for the treatment of diabetic wound infections . Meta-analyses of such studies indicate that stem cell mobilization in these clinical conditions is safe and potentially effective in improving surrogate outcome measures and hard endpoints (such as rates of wound healing and amputation).

This study plans to evaluate whether a single injection of Plerixafor improves wound healing in diabetic patients with stage III-IV (neuro)ischemic wounds.

DETAILED DESCRIPTION:
Chronic non-healing wounds represent a major source of morbidity, disability, and mortality in diabetic patients. Diabetes is the leading cause of non-traumatic limb amputations worldwide. Many patients with ischemic or neuroischemic wounds are not candidate to surgical/endovascular revascularization, owing to anatomical vascular reasons or for the underlying conditions and co-morbidities. Therefore, identification of novel medical treatment strategies to improve wound healing in diabetic patients is a major challenge for clinicians, researchers, and health care systems.

Defects in bone marrow (BM)-derive stem and progenitor cells, including EPCs, contribute to diabetic complications. Stem cell mobilizing agents have been previously studied as an adjunctive therapy for critical limb ischemia and chronic non-healing wounds in diabetic and non-diabetic patients, as well as for the treatment of diabetic wound infections . Meta-analyses of such studies indicate that stem cell mobilization in these clinical conditions is safe and potentially effective in improving surrogate outcome measures and hard endpoints (such as rates of wound healing and amputation).

However, diabetes impairs the response to the most commonly agent used to mobilize stem cells, namely human recombinant granulocyte colony stimulating factor (hrG-CSF). This notion comes from extensive data in animal models, a retrospective case series in patients with hematological disorders, a meta-analysis of studies conducted in patients with cardiovascular disease, and our proof-of-concept prospective study in otherwise healthy outpatients. Vice versa, our data strongly indicate that diabetic patients adequately mobilize stem/progenitor cells (including vascular progenitors, like EPCs) in response to the CXCR4 antagonist Plerixafor. Plerixafor (Mozobil, Sanofi) is clinically available in Europe (including Italy) as a second-line regimen for stem cell mobilization in patients with myeloma or lymphoma scheduled for autotransplantation, only in combination with hrG-CSF, after failure of hrG-CSF alone, to mobilize a sufficient amount of CD34+ stem cells to start apheresis. Preclinical studies in animal models of delayed and diabetic wound healing support the idea that Plerixafor can be effective as an adjunct therapy to accelerate diabetic wound healing.

This study plans to evaluate whether a single injection of Plerixafor improves wound healing in diabetic patients with stage III-IV (neuro)ischemic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes
* Men of 18-85 years or post-menopausal women <85 years of age
* Presence of neuroischemic or ischemic diabetic wound(s) of the leg(s) / foot(s) Texas grade 3 or 4, with or without infection.
* Ability to provide informed consent.

Exclusion Criteria:

* Sepsis
* Dialysis or severe chronic kidney disease (eGFR <20ml/min/1.73 mq)
* Advanced liver disease (defined as cirrhosis or transaminases >3 times ULN)
* Clinically relevant abnormalities in white blood cell counts at baseline.
* Hematologic disorders (lymphoma, myeloma, acute or chronic leukemia, chronic myeloproliferative disorders)
* Known or highly suspected solid cancer
* Women with childbearing potential
* Known hypersensitivity to Mozobil (Plerixafor or its components)
* Inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Wound healing rate | 6 months
  Comparison of wound healing rates in the 2 groups, defined as the complete healing of wounds after 6 months from randomization

SECONDARY OUTCOMES:
Wound size | 6 months
  Comparison of changes in wound size over time (up to 6 months) in the 2 groups.
Oxygen tension | 6 months
  Comparison of changes in TcO2 (transcutaneous oxygen tension) over time (up to 6 months) in the 2 groups.
Perfusion | 6 months
  Comparison of changes in ankle/brachial index over time (up to 6 months) in the 2 groups.
Surgical intervention | 6 months
  Comparison of the rates of surgical intervention (including debridement and amputations) at 6 months in the 2 groups.
Stem cell mobilization | 6 months
  Comparison of CD34+ cell mobilization (ratio of cell level at 6 hour post-Plerixafor administration and baseline) in patients with good versus poor outcomes
Incidence of adverse events and reactions | 6 months
  Comparison in the incidence of adverse events and reactions in the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Fadini, MD PhD, Study Chair — University of Padova
Locations (1):
- University Hospital of Padova, Padua, Italy

REFERENCES:
- [Derived] Albiero M, D'Anna M, Bonora BM, Zuccolotto G, Rosato A, Giorgio M, Iori E, Avogaro A, Fadini GP. Hematopoietic and Nonhematopoietic p66Shc Differentially Regulates Stem Cell Traffic and Vascular Response to Ischemia in Diabetes. Antioxid Redox Signal. 2022 Apr;36(10-12):593-607. doi: 10.1089/ars.2021.0097. Epub 2022 Jan 4. PMID 34538132